CLINICAL TRIAL: NCT05551871
Title: Effects of Usage of Simvastatin in Mild to Moderate Traumatic Brain Injury (TBI) Patients. Could it Make a Difference?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Muhammad Hamdi Taha Muhammad, Principal Investigator , anesthesiology and ICU resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Simvastatin and TBI
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin (Active Comparator): the patient will receive simvastatin 40mg
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): the patient will receive placebo drug
  Interventions: Drug: Placebo drug

INTERVENTIONS:
Drug: Simvastatin — the patient will receive Simvastatin for 7 days
  Arms: Simvastatin
Drug: Placebo drug — the patient will receive Placebo drug for 7 days
  Arms: Placebo

SUMMARY:
Traumatic brain injury (TBI) is a common cause of long-term neurological morbidity, with devastating personal and societal consequences. At present, no pharmacological intervention clearly improves outcomes, and therefore a compelling unmet clinical need remains. 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors, or "statins," offer a potential novel therapeutic strategy for TBI. In this study the investigators will study primarily the effect of statins on 30-day mortality rate which is defined as death within 30 days of TBI presentation where the occurrence of TBI is hour 0 or day 0 and secondarily evaluation of duration of ICU stay associated with or without complications.

DETAILED DESCRIPTION:
TBI is defined as an alteration in brain function, or other evidence of brain pathology, caused by an external force.

[A] Alteration in brain function is defined as 1 of the following clinical signs:

* Any period of loss of or a decreased level of consciousness.
* Any loss of memory for events immediately before (retrograde amnesia) or after the injury (Post traumatic amnesia)
* Neurologic deficits (weakness, loss of balance, change in vision, dyspraxia paresis/plegia [paralysis], sensory loss, aphasia, etc.)
* Any alteration in mental state at the time of the injury (Confusion, disorientation, slowed thinking, etc.) [B] or other evidence of brain pathology: Such evidence may include visual, neuroradiologic, or laboratory confirmation of damage to the brain.

Traumatic brain injury is the most common cause of death and disability in young people.

Traumatic brain injury is graded as mild, moderate, or severe on the basis of the level of consciousness or Glasgow coma scale (GCS) score after resuscitation. Mild traumatic brain injury (GCS 13-15) is in most cases a concussion and there is full neurological recovery, although many of these patients have short-term memory and concentration difficulties. In moderate traumatic brain injury (GCS9-13) the patient is lethargic or stuporous, and in severe injury (GCS 3-8) the patient is comatose, unable to open his or her eyes or follow commands.

The World Health Organization (WHO) estimates that almost 90% of deaths due to injuries occur in low- and middle-income countries (LMICs), where the 85% of population live and this situation will continue to represent an important global health problem in the upcoming years. Of these trauma-related deaths TBI is the main cause of one-third to one-half, and the leading cause of disability under forty years-old (15-20/100,000 populations per year).

One of the most significant disabilities associated with TBI is short- and long-term cognitive deficits. Approximately 65% of patients with moderate to severe TBI report long-term problems with cognitive functioning, and as many as 15% with mild TBI have persistent problems that often include cognitive deficits .These deficits interfere with work and daily living activities, exacting a personal and economic cost that is difficult to quantify. However, despite substantial efforts, few therapeutic options exist to prevent or alleviate cognitive dysfunction after TBI in humans.

The 3-hydroxy-3-methylglutaryl coenzyme A (HMG CoA) reductase inhibitors, also known as "statins," are an ideal candidate therapy for acute brain injury. Statins influence multiple mechanisms of acute and secondary neuronal injury; they have endothelial and vasoactive properties, as well as anti-oxidant, anti-inflammatory, anti-excitotoxicity, and anti-thrombotic effects. Statin treatment would be practical to implement in TBI because Statins have wide availability, Food and Drug Administration approval, a favorable adverse event profile, and a track record of safety in critically ill populations.

CLASSIFICATION OF STATINS All statins contain an HMG-like component that binds to HMG-CoA reductase.other molecular characteristics vary across the class, including potency, lipophilicity, metabolism, and pharmacokinetics. Lovastatin, pravastatin, and simvastatin are obtained from fungi; atorvastatin, rosuvastatin, fluvastatin, and pravastatin are synthetic. Statin potency refers to the degree of HMG-CoA reductase inhibition. Statins are potent inhibitors of cholesterol biosynthesis via HMG-CoA reductase inhibition. Statins are widely used to decrease low-density lipoprotein (LDL) levels and lower the risk of cardiovascular events. As clinical experience with statins has increased, evidence suggests that the cardiovascular benefit may not solely be related to cholesterol lowering, but also to systemic and vascular anti-inflammatory effects. There is growing evidence that statins have additional properties that are neuroprotective, also independent of serum cholesterol effects. The therapeutic effects of statins in brain injury may be divided according to mechanism from most acute to more chronic: acute lesional effects, anti-inflammatory and anti-excitotoxic effects, vascular and endothelial effects, anti-apoptotic effects, and effects on neurogenesis and angiogenesis The statins are inhibitors of cholesterol biosynthesis, and they have additional pleiotropic properties that make them attractive multipotential neuroprotective drugs. Statins increase endothelium-derived nitric oxide production and reduce vascular inflammation, thereby improving the microvasculature after traumatic insult. In in vitro models statins protect cortical neurons from NMDA-induced excitotoxic death , and statin treatment significantly improves neuronal survival following TBI .Statins may also promote the growth and differentiation of new neurons after brain injury , and their ability to increase neurogenesis may be in part due to up regulation of neurotrophic factors (e.g. BDNF) Notably, statins exert powerful anti-inflammatory effects, in part by decreasing the formation of isoprenoids In TBI models, statins have been shown to significantly reduce proinflammatory cytokine production and attenuate microglial activation and cerebral edema formation, while increasing BBB integrity. Experimental studies have shown that statins target multiple secondary injury pathways and significantly improve functional recovery after TBI. Furthermore, the therapeutic window for this class of drugs is relatively large, with treatment 24 h after TBI resulting in long-term functional improvements and reduced neuronal cell loss . As such, statins possess key preclinical neuroprotective characteristics that make them suitable candidates for clinical translation. Importantly, statins have a long clinical track record in critically ill patients; they are easy to administer, are well tolerated and have well-defined side effects . A small prospective, randomized, double-blind clinical trial in TBI has been performed using the statin drug rosuvastatin, and treatment showed modest improvements in TBI associated amnesia and disorientation time outcomes .

ELIGIBILITY:
Inclusion Criteria:

* adult patients from 18 to 40 years old with mild to moderate TBI

Exclusion Criteria:

* immunotherapy
* diabetic
* previous CNs dysfunction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
30-day mortality rate | 30 days
  defined as death within30 days of TBI presentation where the occurrence of TBI is hour 0 or day 0.

SECONDARY OUTCOMES:
1. ICU stay | 30 days
  Days of ICU stay
Complications | 30 days
  convulsions, fever, Infection or wound complications including SSI
Glasgow Coma Scale (GCS) | 30 days
  a clinical scale used to reliably measure a person's level of consciousness after a brain injury. The scale assesses patients according to three aspects of responsiveness: eye-opening, motor, and verbal responses. Reporting each of these separately provides a clear, communicable picture of a patient's state. GCS is evaluated on a scale of 15 where 15 is the highest showing the participant to be responsive and 3 is the lowest on the scale showing the participant to be completely unresponsive.
CBC | 30 days
  Complete Blood Count
CRP | 30 days
  C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Emad Zarief Kamel, MD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Menon DK, Schwab K, Wright DW, Maas AI; Demographics and Clinical Assessment Working Group of the International and Interagency Initiative toward Common Data Elements for Research on Traumatic Brain Injury and Psychological Health. Position statement: definition of traumatic brain injury. Arch Phys Med Rehabil. 2010 Nov;91(11):1637-40. doi: 10.1016/j.apmr.2010.05.017. PMID 21044706
- [Background] Barlow KM. Traumatic brain injury. Handb Clin Neurol. 2013;112:891-904. doi: 10.1016/B978-0-444-52910-7.00011-8. PMID 23622299
- [Background] Iaccarino C, Carretta A, Nicolosi F, Morselli C. Epidemiology of severe traumatic brain injury. J Neurosurg Sci. 2018 Oct;62(5):535-541. doi: 10.23736/S0390-5616.18.04532-0. PMID 30182649
- [Background] Peng W, Yang J, Yang B, Wang L, Xiong XG, Liang Q. Impact of statins on cognitive deficits in adult male rodents after traumatic brain injury: a systematic review. Biomed Res Int. 2014;2014:261409. doi: 10.1155/2014/261409. Epub 2014 Jul 23. PMID 25157352
- [Background] Wible EF, Laskowitz DT. Statins in traumatic brain injury. Neurotherapeutics. 2010 Jan;7(1):62-73. doi: 10.1016/j.nurt.2009.11.003. PMID 20129498
- [Background] Kumar A, Loane DJ. Neuroinflammation after traumatic brain injury: opportunities for therapeutic intervention. Brain Behav Immun. 2012 Nov;26(8):1191-201. doi: 10.1016/j.bbi.2012.06.008. Epub 2012 Jun 21. PMID 22728326